CLINICAL TRIAL: NCT05637879
Title: Randomized Controlled Trial of Glecaprevir/Pibrentasvir for the Treatment of Post-traumatic Stress Disorder
Brief Title: Glecaprevir/Pibrentasvir for Post-traumatic Stress Disorder
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bradley Watts, Staff Psychiatrist, White River Junction Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1698661; W81XWH22C0147 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-11-15; First posted 2022-12-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-08

CONDITIONS: PTSD
Keywords: PTSD; Antiviral; Hepatitis C
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Hepatitis C | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Intervention Model Description: Blinded placebo-controlled randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Drug (Active Comparator): Glecaprevir 100 mg/Pibrentasvir 40 mg, 3 oral tablets once daily for 8 weeks.
  Interventions: Drug: Glecaprevir/pibrentasvir
- Placebo (Placebo Comparator): Placebo, 3 oral tablets once daily for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glecaprevir/pibrentasvir — Direct-acting antiviral, Food & Drug Administration (FDA) approved for the treatment of hepatitis C viral infection
  Other Names: Mavyret
  Arms: Active Drug
Other: Placebo — Compounded, inactive pill equal in appearance to active study drug
  Arms: Placebo

SUMMARY:
A double-blind randomized placebo-controlled trial to further investigate glecaprevir/pibrentasvir (GLE/PIB), a direct acting antiviral (DAA) that has been associated with posttraumatic stress disorder (PTSD) symptom improvement when prescribed for the treatment of chronic hepatitis C viral infection (HCV).

DETAILED DESCRIPTION:
N=92 patients with posttraumatic stress disorder (PTSD) will be enrolled into a double-blind randomized placebo-controlled trial to further investigate glecaprevir/pibrentasvir (GLE/PIB), a direct acting antiviral (DAA) that has been associated with PTSD symptom improvement when prescribed for the treatment of chronic hepatitis C viral infection (HCV). The research is intended to test the efficacy of GLE/PIB for PTSD symptom improvement in the absence of HCV.

Primary Aims:

Aim 1: Determine the efficacy of GLE/PIB for PTSD symptom improvement. Aim 2: Determine the efficacy of GLE/PIB for functioning improvement among patients with PTSD.

Aim 3: Assess the safety and tolerability of GLE/PIB treatment for patients with PTSD in the absence of HCV.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-70 years
2. Weight ≥ 45 kg
3. Diagnosed with PTSD as determined by the CAPS-5 within seven days of enrollment
4. Eligible for Veterans Affairs healthcare
5. If person with childbearing potential, use of acceptable method of birth control (i.e., effective contraceptives, abstinence) is required.
6. Able to read, understand, and sign the informed consent document.

Exclusion (unable to participate) Criteria:

1. Pregnant or lactating person
2. Moderate or severe hepatic impairment (Child-Pugh B or C)
3. History of prior hepatic decompensation
4. Current use of drugs listed as having significant drug interactions on prescribing label
5. Advanced liver disease
6. Current or prior hepatitis B infection
7. Prior clinical use of GLE/PIB or HCV NS5A inhibitor AND NS3/4A protease inhibitor
8. Current HCV infection
9. Current psychosis or mania
10. Significant suicidal ideation
11. Unstable medical conditions
12. Current severe alcohol or substance use disorder (excluding nicotine)
13. Evidence-based PTSD psychotherapy changes in the past two months
14. Evidence-based PTSD medication changes in the past two months

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Administered Post-Traumatic Stress Disorder Scale version 5 (CAPS-5) | Change from Baseline CAPS score at 8 weeks
  Queries the frequency and intensity of symptoms of post-traumatic stress disorder (PTSD). The score ranges from 0-80 with a higher score indicating worse symptoms. It is considered the gold standard for diagnosis and symptoms assessment in PTSD clinical studies.

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Schedule, version 2.0 (WHODAS) | Change from Baseline WHODAS score at 8 weeks
  A 36 item self-report instrument that assesses disability and function across six domains: communicating, getting around, self-care, getting along with people, life activities, and participation in society. The WHODAS has been used as an outcome of function and disability across many disorders and is commonly used in mental health treatment trials. The total score ranges from 0-180 with a higher score indicating worse functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley V Watts, MD, MPH, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- White River Junction VAMC, White River Junction, Vermont, United States

IPD SHARING:
Plan to Share IPD: No